CLINICAL TRIAL: NCT03518125
Title: Randomized, Active-Comparison, Double-Blind, Phase 2 Study to Assess the Safety and Immunogenicity of Anthrax Vaccine Adsorbed (BioThrax®) Without and With CPG 7909 Adjuvant (AV7909 Anthrax Vaccine), Using a Post-Exposure Prophylaxis Dosing Regimen in Adults 66 Years of Age or Older in Stable Health in Comparison to Adults 18-50 Years of Age in Stable Health
Brief Title: BARDA Securing Anthrax Immunity For the Elderly
Acronym: B-SAFE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Collaborators: Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BP-C-17001; HHSO100201400004I (Other Grant/Funding Number: BARDA)
Record Dates: First submitted 2018-04-24; First posted 2018-05-08 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Anthrax
Keywords: Anthrax; Bacillaceae Infections; Gram-Positive Bacterial Infections; Bacterial Infections; Anthrax Vaccine Adsorbed; BioThrax; AV7909; CPG 7909; Adjuvant; Vaccines; Post-exposure Prophylaxis
MeSH Terms: conditions — Anthrax; Bacillaceae Infections; Gram-Positive Bacterial Infections; Bacterial Infections | interventions — Biothrax

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either BioThrax or AV7909. Randomization will be stratified by sex and age (18-50, 66-74, and ≥75 years). Subjects ≥66 years of age will be randomized 1:1:1:1 within stratum across 4 treatment arms (approximately 50 subjects per group), and subjects 18 through 50 years of age will be randomized 1:1 within stratum across 2 treatment arms (approximately 50 subjects per group). Once randomized, subjects will receive 3 vaccinations, each separated by approximately 14 days, on Day 1, Day 15, and Day 29, based on their assigned treatment arm.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Age ≥ 66, BioThrax (Days 1, 15, 29) (Experimental): Subjects dosed on Days 1, 15, and 29 with 0.5 mL BioThrax.
  Interventions: Biological: BioThrax
- Age ≥ 66, AV7909 (Days 1, 15, 29) (Experimental): Subjects dosed on Days 1, 15, and 29 with 0.5 mL AV7909.
  Interventions: Biological: AV7909
- Age ≥ 66, AV7909 (Days 1 and 15) (Experimental): Subjects dosed on Days 1 and 15 with 0.5 mL AV7909 and on Day 29 with 0.5 mL placebo.
  Interventions: Biological: AV7909; Drug: Sodium chloride injection USP, 0.9% (placebo)
- Age ≥ 66, AV7909 (Days 1 and 29) (Experimental): Subjects dosed on Days 1 and 29 with 0.5 mL AV7909 and on Day 15 with 0.5 mL placebo.
  Interventions: Biological: AV7909; Drug: Sodium chloride injection USP, 0.9% (placebo)
- Age18-50, BioThrax (Days 1, 15, 29) (Active Comparator): Subjects dosed on Days 1, 15, and 29 with 0.5 mL BioThrax.
  Interventions: Biological: BioThrax
- Age 18-50, AV7909 (Days 1 and 15) (Active Comparator): Subjects dosed on Days 1 and 15 with 0.5 mL AV7909 and on Day 29 with 0.5 mL placebo.
  Interventions: Biological: AV7909; Drug: Sodium chloride injection USP, 0.9% (placebo)

INTERVENTIONS:
Biological: BioThrax — Other Names:
  Anthrax Vaccine Adsorbed (AVA)
  Arms: Age ≥ 66, BioThrax (Days 1, 15, 29); Age18-50, BioThrax (Days 1, 15, 29)
Biological: AV7909 — Anthrax Vaccine Absorbed plus CPG 7909 Adjuvant
  Other Names: AV7909 Anthrax Vaccine Adsorbed; NuThrax
  Arms: Age 18-50, AV7909 (Days 1 and 15); Age ≥ 66, AV7909 (Days 1 and 15); Age ≥ 66, AV7909 (Days 1 and 29); Age ≥ 66, AV7909 (Days 1, 15, 29)
Drug: Sodium chloride injection USP, 0.9% (placebo) — Other Names:
  Saline Solution
  Arms: Age 18-50, AV7909 (Days 1 and 15); Age ≥ 66, AV7909 (Days 1 and 15); Age ≥ 66, AV7909 (Days 1 and 29)

SUMMARY:
This study is designed to assess the safety and ability of BioThrax and AV7909 anthrax vaccines to generate an immune response in adults ≥ 66 years of age in stable health in comparison to adults 18-50 years of age in stable health.

DETAILED DESCRIPTION:
This is a phase 2, randomized, active-controlled, double-blinded, multi-site study to assess the safety and immunogenicity of BioThrax (Anthrax Vaccine Adsorbed) and AV7909 (Anthrax Vaccine Adsorbed plus CPG 7909 adjuvant) using a post-exposure prophylaxis dosing regimen in adults ≥ 66 years of age in stable health. The safety and immunogenicity profile of BioThrax and AV7909 in adults ≥ 66 years of age will also be compared to the safety and immunogenicity profile of subjects 18-50 years of age in stable health. The main study goal is to determine optimal dosing for AV7909 in the elderly population. Subjects will receive either 3 doses of BioThrax, 3 doses of AV7909, or 2 doses of AV7909 and 1 dose of placebo. Doses will be administered approximately 14 days apart. Subjects will be followed for safety assessment for 12 months following the last dose. The expected study duration is approximately 14 months per subject.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant females, 66 years of age or older at the time of randomization for the elderly population, or 18 through 50 years of age at the time of randomization for the younger population.
2. Females who are of childbearing potential and are sexually active with a male partner must agree to use an acceptable method of birth control from Screening to Day 64 and must have used a reliable birth control method for at least 2 months prior to Screening.

   1. A female of childbearing potential is defined as post onset menarche and pre-menopausal female capable of becoming pregnant. This does not include females who meet any of the following conditions: menopausal >2 years, tubal ligation >1 year, bilateral salpingo-oophorectomy, or hysterectomy.
   2. Adequate contraception is defined as a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label. Examples include: oral contraceptives, either combined or progestogen alone; injectable progestogen; implants of etenogestrel or levonorgestrel; estrogenic vaginal ring; percutaneous contraceptive patches; intrauterine device or intrauterine system; male partner sterilization at least 6 months prior to the female subject's Screening Visit, and this male is the sole partner for that subject (the information on the male partner's sterility can come from the site personnel's review of the subject's medical records or interview with the subject on her medical history); male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository); male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository).
3. Able to provide written informed consent prior to initiation of any study procedures. As part of the consent process, subjects must be able to demonstrate understanding by passing the "Assessment of Understanding Questionnaire" within 2 attempts. Passing is defined as being able to answer all questions correctly.
4. In relatively stable health based on site investigator's judgment, as determined by medical history, physical examination, and the following criteria:

   1. Stable health for age (defined as no new conditions per medical history, new medications in a different therapeutic class, or change in daily dose of existing prescription medications within the 45 days preceding Screening). Effective treatment (to resolution) of an acute infection (e.g., urinary tract infection, cellulitis, otitis, or bronchitis) with an antibiotic within 45 days preceding Screening will not be considered a deviation from this inclusion criterion as long as the antibiotic therapy was completed at least one week prior to Screening and no signs or symptoms of the infection have been present since the completion of treatment. Any prescription change that is due to change of health care provider or insurance company, or that is made for reasons that do not reflect a change in disease status (e.g., financial considerations), as long as within the same general class of medication, will not be considered a deviation from this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site investigator, will not be considered a deviation from this inclusion criterion.
   2. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site investigator, these pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and their use is not for management of a worsening of medical diagnosis or condition. Note: Topical, nasal, and inhaled medications (with the exception of steroids, as outlined in the subject exclusion criteria) and vitamins are permitted.
5. Have a body mass index (BMI) less than 35.0 kg/m2 at Screening. (BMI will not be reassessed prior to subsequent vaccinations.)
6. Have access to a consistent and reliable means of telephone contact, which may be home, workplace, or by personal mobile electronic device.
7. Are available and able to comply with all study visits.

Exclusion Criteria:

1. Females who have a positive urine pregnancy test at Screening or within 24 hours prior to each study vaccination or women who are breastfeeding.
2. Have a requirement for skilled nursing care.
3. Have a history of severe reactions to components of AVA or CPG 7909, e.g., formaldehyde, benzethonium chloride (phemerol), or aluminum.
4. Have a history of latex sensitivity.
5. Have a history of ever receiving a vaccine for anthrax prior to Screening, or had an anthrax infection.
6. Have any medical, psychiatric, or social condition that, in the opinion of the site investigator, unfavorably alters the risk-benefit of subject participation, or is likely to interfere with study compliance or assessments, or is likely to confound interpretation of safety or immunogenicity data.
7. Have any diagnosis, current or past, of a potentially immune-mediated medical condition, such as Guillain-Barré syndrome, narcolepsy, or an autoimmune or chronic inflammatory disease.
8. Have any diagnosis, current or past, of schizophrenia or bipolar disorder.
9. Have been hospitalized for psychiatric illness, have a history of suicide attempt, or confinement for danger to self or others within the preceding 10 years prior to Screening and each study vaccination.
10. Have a history of alcohol or drug abuse (per investigator's judgment) within 5 years prior to Screening and each study vaccination, or test positive for drugs of abuse at Screening (including for cannabis, even where legal). Benzodiazepines for anxiety disorders and stimulants for attention deficit hyperactivity disorder are not exclusionary if the subject has been on a stable dose for more than 3 months prior to Screening and each study vaccination and if the subject can produce a valid, current prescription for the medication. Propoxyphene, opioids, or combinations containing these medications (including as used for opioid addiction) are not permitted regardless of prescription status. Note: A positive Screening urine drug screen may not be repeated. (Drug screen will not be repeated prior to subsequent vaccinations.)
11. Have known human immunodeficiency virus (HIV), or acute or chronic hepatitis B or hepatitis C infection based on medical history; or test positive for any of these at Screening. Subjects who have been effectively treated for hepatitis C, as evidenced by a negative hepatitis C ribonucleic acid (RNA) confirmation test and who no longer require antiviral therapy, are eligible for participation. (Screening tests will not be repeated prior to subsequent vaccinations.)
12. Have known active neoplastic disease or a history of any hematologic malignancy. However, subjects with superficial skin cancer who do not require intervention other than local excision are not excluded.
13. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy (cytotoxic) or radiation therapy within 3 years prior to Screening and each study vaccination.
14. Have taken any systemic immunosuppressive agents, including immunomodulators, 6 months prior to Screening and each study vaccination. Allergen immunotherapy (desensitization) is not exclusionary. Allergen immunotherapy (desensitization) does not include systemic antibodies such as benralizumab, mepolizumab, or omalizumab; these are exclusionary.
15. Are suffering from or have a history of neuralgia, paresthesia, or neuritis within 90 days prior to Screening and each study vaccination; or have any history of stroke.
16. Have had convulsions or encephalomyelitis within three years prior to Screening and each study vaccination.
17. Have received immunoglobulin or other blood products (with the exception of Rho[D] immune globulin) within 90 days prior to Screening and each study vaccination.
18. Have received an experimental agent within 180 days prior to the first study vaccination, or expects to participate in another clinical trial with an interventional agent during the study period. This includes licensed or unlicensed vaccines, drugs, biologics, devices, blood products, or medications. Participation in an observational study is not exclusionary as long as it doesn't interfere with study visits or procedures (e.g., blood collection volume restrictions).
19. Have taken oral or parenteral corticosteroids of any dose within 30 days prior to each study vaccination.
20. Have taken high-dose inhaled corticosteroids within 30 days prior to each study vaccination. High-dose is defined as >800 mcg/day of beclomethasone dipropionate or equivalent. Lower doses of inhaled corticosteroids are not exclusionary.
21. Have received any licensed live vaccine within 30 days prior to the first study vaccination or planned receipt from the first study vaccination through Visit 10 (Day 64).
22. Have received any licensed inactivated vaccine within 14 days prior to the first study vaccination or planned receipt from the first study vaccination through Visit 10 (Day 64).
23. Have an acute illness, as determined by the site investigator, within 72 hours prior to each study vaccination.

    1. If subject's oral temperature is above 100.0°F (37.8°C), the subject may be re-assessed for eligibility within the visit window (+3 Days).
    2. An acute illness that is nearly resolved, with only minor residual symptoms remaining, is allowable if, in the opinion of the site investigator, the residual symptoms will not interfere with the ability of study staff to assess safety parameters as required by the protocol.
    3. For bacterial infections that have been successfully treated with antibiotics, inclusion criterion 4a applies.
24. Have a history of myocardial infarction or ischemia, or have electrocardiogram (ECG) findings of myocardial infarction, ischemia, strain, complete bundle branch block, or ventricular arrhythmias (other than unifocal premature ventricular contractions ≤2/minute). Additionally, other cardiac history or ECG findings, which in the opinion of the investigator represent a potentially unstable or unacceptably high risk of an adverse cardiac outcome, are exclusionary. (ECG will not be repeated prior to subsequent vaccinations.)
25. Have any laboratory test result or clinical findings (including vital signs) that singly or in combination are, in the investigator's opinion, likely to unfavorably alter the risk-benefit of subject participation or to confound study safety or immunogenicity results. Additionally, the following are exclusionary:

    1. Any clinically significant Grade 3 laboratory or vital sign result, or any Grade 4 laboratory or vital sign result (regardless of assessed significance) at Screening. For subsequent vaccinations, abnormal laboratory results and vital sign results postvaccination will be assessed against the rules for early termination of dosing.
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 times the upper limit of normal (ULN), or bilirubin >1.5 times the ULN unless isolated Gilbert's syndrome.
    3. Creatinine >1.5 times ULN for age and sex.
    4. White blood cell count <3,000/μL or >12,500/μL; absolute neutrophil count <1200/μL; absolute lymphocyte count <750/μL; hemoglobin <10 g/dL females, or <11.5 g/dL males; platelet count <75,000/μL.
    5. Hemoglobin A1C (HbA1C) >7.0% at Screening. (HbA1C will not be repeated prior to subsequent vaccinations.)

Subjects cannot be rescreened for exclusionary laboratory test results. Potentially exclusionary vital sign results may be repeated, but unless they have resolved to a Grade 3 designation or less and are not considered clinically significant, the subject should be excluded. The most recent laboratory and vital sign results will be used when determining eligibility for subsequent vaccinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Fierro, MD, Principal Investigator — Johnson County Clin-Trials; Derek Muse, MD, Principal Investigator — JBR Clinical Research; Stephan Sharp, MD, Principal Investigator — Clinical Research Associates, Inc.; Cynthia Strout, MD, Principal Investigator — Coastal Carolina Research Center
Locations (4):
- United States (4):
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolfe DN, Espeland EM, Gao Y, Lu D, Blatner G, Amass K, Horwith G, Tong XM, Hopkins R, David GL, Jepson BM, King JC Jr. Evaluation of BioThrax(R) and AV7909 anthrax vaccines in adults 66 years of age or older. Vaccine. 2020 Nov 25;38(50):7970-7976. doi: 10.1016/j.vaccine.2020.10.053. Epub 2020 Oct 28. PMID 33129609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 469 participants were screened at 4 sites in the US between May 14, 2018 - November 8, 2018, of which 305 were randomized and vaccinated between May 17, 2018 - November 12, 2018.
Groups:
- Age ≥ 66 Years: BioThrax (Day 1, Day 15, and Day 29); Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29): Participants dosed subcutaneously (SC) on Days 1, 15, and 29 with 0.5 mL BioThrax
- Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29): Participants dosed intramuscularly (IM) on Days 1, 15, and 29 with 0.5 mL AV7909
- Age ≥ 66 Years: AV7909 (Days 1, Day 15) With Placebo (Day 29); Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29): Participants dosed intramuscularly (IM) on Days 1 and 15 with 0.5 mL AV7909 and dosed IM on Day 29 with 0.5 mL placebo
- Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15): Participants dosed intramuscularly (IM) on Days 1 and 29 with 0.5 mL AV7909 and dosed IM on Day 15 with 0.5 mL placebo
Period: Overall Study
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, and Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Days 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Started | 50 | 50 | 49 | 52 | 52 | 52
Completed | 48 | 46 | 49 | 51 | 48 | 44
Not Completed | 2 | 4 | 0 | 1 | 4 | 8
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 3 | 5
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 1 | 3
Not completed — Missed Day 394 Visit | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population includes all randomized participants who received any amount of study vaccination.
Groups:
- Age ≥ 66 Years: BioThrax (Day1, Day 15, Day 29); Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29): Participants dosed subcutaneously (SC) on Days 1, 15, and 29 with 0.5 mL BioThrax
- Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29); Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29): Participants dosed intramuscularly (IM) on Days 1 and 15 with 0.5 mL AV7909 and dosed IM on Day 29 with 0.5 mL placebo
- Total: Total of all reporting groups
Arm/Group | Age ≥ 66 Years: BioThrax (Day1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Total
Number analyzed (Participants) | 50 | 50 | 49 | 52 | 52 | 52 | 305
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 51 | 51 | 102
  >=65 years | 50 | 50 | 49 | 52 | 0 | 0 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (5.89) | 71.2 (4.76) | 72.8 (4.88) | 72.5 (5.04) | 33.5 (9.46) | 33.7 (9.55) | 59.1 (19.63)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 28 | 29 | 27 | 31 | 29 | 29 | 173
  Gender: Male | 22 | 21 | 22 | 21 | 23 | 23 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 1 | 0 | 3 | 7
  Not Hispanic or Latino | 49 | 48 | 48 | 50 | 51 | 48 | 294
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 2 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 3 | 2 | 6 | 3 | 20
  White | 46 | 46 | 46 | 47 | 45 | 47 | 277
  More than one race | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 49 | 52 | 52 | 52 | 305

OUTCOME MEASURES:

1. Primary Outcome: Solicited Local Reactogenicity Symptoms
Description: Count of participants who experienced at least one of the following during the time frame specified on the arm which received the vaccination: injection site warmth, tenderness, itching, pain, restriction of range of arm motion, erythema/redness, palpable or observable lump, induration/swelling, or bruising.
Time Frame: Day 1-8, Day 15-22, Day 29-36 (within 8 days of each vaccination, inclusive of the vaccination day)
Population: Safety population includes all randomized participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≥ 66 Years: BioThrax (Day1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 50 | 50 | 49 | 52 | 52 | 52
Participants | 46 | 43 | 40 | 45 | 50 | 50

2. Primary Outcome: Solicited Systemic Reactogenicity Symptoms
Description: Count of participants who experienced at least one of the following during the time frame specified on the arm which received the vaccination: fatigue, myalgia/muscle ache, headache, and fever.
Time Frame: Day 1-8, Day 15-22, Day 29-36 (within 8 days of each vaccination, inclusive of the vaccination day)
Population: Safety population includes all randomized participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29); Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29): Participants dosed subcutaneously (SC) on Days 1, 15, and 29 with 0.5 mL BioThrax
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 50 | 50 | 49 | 52 | 52 | 52
Participants | 14 | 23 | 18 | 20 | 15 | 35

3. Primary Outcome: Seroprotection Based on Toxin Neutralization Antibody (TNA) 50% Neutralization Factor (NF50) Antibody Level, Defined as a TNA NF50 Antibody Level ≥0.56
Description: The percentage of participants achieving seroprotection based on TNA NF50. A 70% probability of survival was associated with a TNA NF50 level of 0.56 in rabbits exposed to Bacillus anthracis, the bacteria that causes anthrax.
Time Frame: Day 64
Population: Immunogenicity per protocol population (IPPP) includes all randomized participants who received a full dose of the correct vaccine at Days 1, 15, and 29 within the protocol specified windows, had determinate assay results at Day 64 (within window), and had no major protocol deviations that may have impacted immunogenicity assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 41 | 39 | 41 | 41 | 42 | 38
Participants | 7 | 37 | 19 | 40 | 22 | 23

4. Secondary Outcome: Treatment-emergent Unsolicited Adverse Events (AEs)
Description: The count of participants who experienced at least one post-vaccination unsolicited AE (i.e. AEs not included in the solicited local and systemic adverse event list through Day 50 and those reported as a serious AE, medically attended adverse event (MAAE), or potentially immune-mediated medical condition (PIMMC) after Day 50).
Time Frame: Day 1 through Day 394
Population: Safety population includes all randomized participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 50 | 50 | 49 | 52 | 52 | 52
Participants | 41 | 34 | 32 | 39 | 30 | 26

5. Secondary Outcome: Treatment-emergent Serious Adverse Events (SAEs)
Description: The count of participants who experienced at least one post-vaccination SAE
Time Frame: Day 1 through Day 394
Population: Safety population includes all randomized participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 50 | 50 | 49 | 52 | 52 | 52
Participants | 1 | 3 | 3 | 2 | 0 | 2

6. Secondary Outcome: Treatment-emergent Medically Attended Adverse Events (MAAEs)
Description: Count of participants who experienced at least one adverse event that requires a visit to medical personnel, including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason occurring post-vaccination.
Time Frame: Day 1 through Day 394
Population: Safety population includes all randomized participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 50 | 50 | 49 | 52 | 52 | 52
Participants | 27 | 23 | 21 | 23 | 13 | 14

7. Secondary Outcome: Treatment-emergent Potentially Immune Mediated Medical Conditions (PIMMCs)
Description: Count of participants who experienced at least one medical condition that was potentially immune mediated occurring post-vaccination
Time Frame: Day 1 through Day 394
Population: Safety population includes all randomized participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 50 | 50 | 49 | 52 | 52 | 52
Participants | 0 | 0 | 1 | 0 | 0 | 0

8. Secondary Outcome: Solicited Local Reactogenicity Symptoms on the Contralateral Arm
Description: Count of participants who experienced at least one of the following during the time frame specified on the arm which did not receive the vaccination: injection site warmth, tenderness, itching, pain, restriction of range of arm motion, erythema/redness, palpable or observable lump, induration/swelling, or bruising.
Time Frame: Day 1-8, Day 15-22, Day 29-36 (within 8 days of each vaccination, inclusive of the vaccination day)
Population: Safety population includes all randomized participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 50 | 50 | 49 | 52 | 52 | 52
Participants | 11 | 6 | 3 | 5 | 7 | 2

9. Secondary Outcome: TNA NF50 Antibody Levels
Description: A higher TNA NF50 antibody level means a better immune response to the vaccine.
Time Frame: Days 1, 8, 22, 29, 36, 43, 50, 64, 85, 181, and 394
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 41 | 39 | 41 | 41 | 42 | 38
Titers
  Day 1 | .03 [.03 to .03] | .03 [.03 to .03] | .03 [.03 to .03] | .03 [.03 to .03] | .03 [.03 to .03] | .03 [.03 to .03]
  Day 8 | .03 [.03 to .03] | .03 [.03 to .03] | .03 [.03 to .03] | .03 [.03 to .03] | .03 [.03 to .04] | .03 [.03 to .03]
  Day 22 | .04 [.03 to .05] | .25 [.14 to .45] | .23 [.14 to .39] | .10 [.07 to .14] | .08 [.05 to .11] | .67 [.48 to .95]
  Day 29 | .11 [.07 to .16] | .77 [.49 to 1.20] | .80 [.54 to 1.17] | .12 [.08 to .16] | .43 [.30 to .63] | 1.02 [.80 to 1.31]
  Day 36 | .36 [.25 to .52] | 2.92 [1.90 to 4.48] | .75 [.50 to 1.11] | 2.98 [2.08 to 4.27] | .84 [.60 to 1.16] | 1.06 [.82 to 1.38]
  Day 43 | .55 [.45 to .68] | 4.26 [3.20 to 5.66] | .69 [.47 to 1.02] | 6.73 [5.19 to 8.72] | .94 [.73 to 1.21] | .94 [.72 to 1.21]
  Day 50 | .45 [.36 to .56] | 3.38 [2.58 to 4.43] | .60 [.41 to .88] | 5.30 [4.12 to 6.81] | .79 [.61 to 1.03] | .84 [.64 to 1.10]
  Day 64 | .32 [.25 to .41] | 2.36 [1.83 to 3.06] | .44 [.29 to .64] | 3.42 [2.63 to 4.43] | .59 [.45 to .78] | .69 [.53 to .89]
  Day 85 | .20 [.15 to .26] | 1.48 [1.17 to 1.87] | .30 [.20 to .45] | 2.08 [1.59 to 2.71] | .42 [.30 to .59] | .53 [.40 to .70]
  Day 181 | .05 [.04 to .07] | .37 [.28 to .48] | .12 [.09 to .17] | .34 [.24 to .46] | .12 [.08 to .16] | .23 [.17 to .32]
  Day 394 | .04 [.03 to .04] | .14 [.10 to .20] | .10 [.07 to .13] | .09 [.07 to .12] | .05 [.04 to .07] | .16 [.11 to .23]

10. Secondary Outcome: TNA Effective Dilution Resulting in 50% Neutralization (ED50) Antibody Levels
Description: A higher TNA ED50 antibody level means a better immune response to the vaccine.
Time Frame: Days 1, 8, 22, 29, 36, 43, 50, 64, 85, 181, and 394
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 41 | 39 | 41 | 41 | 42 | 38
Titers
  Day 1 | 16.5 [16.5 to 16.5] | 16.5 [16.5 to 16.5] | 16.5 [16.5 to 16.5] | 16.5 [16.5 to 16.5] | 16.5 [16.5 to 16.5] | 16.5 [16.5 to 16.5]
  Day 8 | 16.5 [16.5 to 16.5] | 16.5 [16.5 to 16.5] | 16.5 [16.5 to 16.5] | 16.5 [16.5 to 16.5] | 17.18 [15.83 to 18.66] | 16.5 [16.5 to 16.5]
  Day 22 | 20.13 [16.84 to 24.06] | 136.20 [77.04 to 240.78] | 122.26 [73.04 to 204.66] | 52.24 [35.89 to 76.03] | 35.66 [24.05 to 52.87] | 322.78 [228.43 to 456.10]
  Day 29 | 54.88 [36.12 to 83.36] | 410.47 [263.48 to 639.47] | 411.94 [280.68 to 604.59] | 63.02 [44.68 to 88.88] | 208.90 [144.37 to 302.28] | 501.88 [391.96 to 642.64]
  Day 36 | 187.97 [130.74 to 270.25] | 1557.95 [1030.38 to 2355.64] | 389.79 [262.37 to 579.07] | 1548.57 [1102.91 to 2174.32] | 410.11 [297.17 to 565.97] | 519.81 [397.84 to 679.18]
  Day 43 | 299.59 [243.47 to 368.64] | 2135.14 [1605.51 to 2839.48] | 361.30 [245.67 to 531.35] | 3490.12 [2737.94 to 4448.95] | 495.07 [386.91 to 633.48] | 497.77 [384.03 to 645.20]
  Day 50 | 250.88 [201.26 to 312.73] | 1658.94 [1265.22 to 2175.19] | 315.10 [214.65 to 462.54] | 2600.22 [2035.57 to 3321.51] | 414.59 [317.69 to 541.06] | 435.56 [331.22 to 572.77]
  Day 64 | 184.31 [145.92 to 232.80] | 1240.66 [976.70 to 1575.97] | 248.04 [168.46 to 365.21] | 1771.46 [1386.67 to 2263.02] | 321.15 [241.54 to 427.00] | 363.05 [279.48 to 471.62]
  Day 85 | 85.20 [63.60 to 114.11] | 650.14 [511.93 to 825.65] | 136.72 [93.76 to 199.38] | 902.39 [689.72 to 1180.63] | 181.14 [130.24 to 251.92] | 224.09 [171.05 to 293.57]
  Day 181 | 25.55 [20.08 to 32.51] | 163.46 [124.59 to 214.46] | 55.87 [40.37 to 77.31] | 151.24 [111.24 to 205.61] | 55.17 [39.33 to 77.39] | 108.67 [80.46 to 146.78]
  Day 394 | 18.29 [16.52 to 20.24] | 74.48 [52.50 to 105.68] | 49.63 [35.44 to 69.49] | 50.29 [37.22 to 67.97] | 27.46 [20.16 to 37.39] | 76.66 [52.84 to 111.21]

11. Secondary Outcome: Enzyme-linked Immunosorbent Assay (ELISA) Anti-protective Antigen (Anti-PA) Immunoglobulin G (IgG) Antibody Levels
Description: A higher ELISA anti-PA IgG antibody level means a better immune response to the vaccine.
Time Frame: Days 1, 8, 22, 29, 36, 43, 50, 64, 85, 181, and 394
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 41 | 39 | 41 | 41 | 42 | 38
Titers
  Day 1 | 4.64 [4.64 to 4.64] | 4.78 [4.49 to 5.09] | 4.64 [4.64 to 4.64] | 4.91 [4.51 to 5.34] | 4.64 [4.64 to 4.64] | 4.64 [4.64 to 4.64]
  Day 8 | 4.64 [4.64 to 4.64] | 4.77 [4.50 to 5.07] | 4.64 [4.64 to 4.64] | 4.96 [4.49 to 5.48] | 4.78 [4.49 to 5.09] | 4.64 [4.64 to 4.64]
  Day 22 | 6.06 [4.78 to 7.68] | 37.28 [22.32 to 62.27] | 40.33 [25.68 to 63.36] | 10.26 [7.19 to 14.62] | 19.61 [12.91 to 29.77] | 80.66 [58.31 to 111.57]
  Day 29 | 29.84 [19.12 to 46.58] | 124.04 [84.60 to 181.85] | 138.17 [97.23 to 196.34] | 11.98 [8.29 to 17.31] | 106.64 [75.80 to 150.02] | 139.82 [112.50 to 173.79]
  Day 36 | 75.98 [52.39 to 110.20] | 347.86 [243.34 to 497.29] | 134.15 [94.10 to 191.25] | 232.20 [165.79 to 325.21] | 180.58 [131.55 to 247.90] | 135.86 [109.84 to 168.05]
  Day 43 | 118.55 [91.81 to 153.09] | 493.50 [382.46 to 636.78] | 122.18 [87.02 to 171.55] | 504.56 [394.48 to 645.35] | 211.41 [164.67 to 271.43] | 120.44 [96.47 to 150.36]
  Day 50 | 100.39 [77.25 to 130.45] | 417.04 [323.71 to 537.28] | 104.99 [74.97 to 147.03] | 418.50 [330.55 to 529.85] | 170.18 [131.18 to 220.79] | 107.84 [86.93 to 133.77]
  Day 64 | 69.71 [53.58 to 90.70] | 334.57 [259.73 to 430.97] | 80.74 [58.90 to 110.69] | 312.36 [246.20 to 396.30] | 124.79 [95.68 to 162.77] | 81.47 [65.02 to 102.08]
  Day 85 | 43.50 [33.31 to 56.82] | 208.58 [162.53 to 267.69] | 48.40 [35.84 to 65.36] | 195.23 [154.55 to 246.62] | 67.78 [51.26 to 89.63] | 50.33 [40.58 to 62.43]
  Day 181 | 9.43 [7.16 to 12.42] | 42.60 [32.44 to 55.92] | 11.70 [8.86 to 15.44] | 36.95 [28.22 to 48.37] | 17.43 [12.76 to 23.81] | 17.90 [13.83 to 23.16]
  Day 394 | 4.76 [4.51 to 5.02] | 12.52 [9.09 to 17.23] | 7.09 [5.74 to 8.76] | 9.24 [7.30 to 11.70] | 6.74 [5.14 to 8.83] | 10.33 [8.17 to 13.06]

12. Secondary Outcome: Seroprotection Based on TNA NF50, Defined as a TNA NF50 Antibody Level ≥0.56
Description: The percentage of participants achieving seroprotection based on TNA NF50 antibody level. A 70% probability of survival was associated with a TNA NF50 level of 0.56 in rabbits exposed to Bacillus anthracis, the bacteria that causes anthrax.
Time Frame: Days 1, 8, 22, 29, 36, 43, 50, 85, 181, and 394
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 41 | 39 | 41 | 41 | 42 | 38
Participants
  Day 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8 | 0 | 0 | 0 | 0 | 0 | 0
  Day 22 | 0 | 18 | 14 | 4 | 2 | 24
  Day 29 | 6 | 27 | 25 | 4 | 18 | 31
  Day 36 | 15 | 35 | 28 | 38 | 33 | 31
  Day 43 | 19 | 37 | 24 | 40 | 33 | 31
  Day 50 | 14 | 38 | 25 | 40 | 30 | 30
  Day 85 | 5 | 34 | 15 | 38 | 13 | 19
  Day 181 | 0 | 11 | 4 | 13 | 2 | 5
  Day 394 | 0 | 3 | 2 | 1 | 1 | 2

13. Secondary Outcome: Seroconversion Based on TNA NF50, Defined as a ≥4-fold Increase Over Pre-vaccination Levels, or a ≥4-fold Increase Over the Lower Limit of Quantification (LLOQ) if the Pre-vaccination Value is Below the LLOQ
Description: The percentage of subjects obtaining seroconversion based on TNA NF50 antibody levels. Seroconversion represents the minimum intended effect of vaccination.
Time Frame: Days 8, 22, 29, 36, 43, 50, 64, 85, 181, and 394
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 41 | 39 | 41 | 41 | 42 | 38
Participants
  Day 8 | 0 | 0 | 0 | 0 | 0 | 0
  Day 22 | 1 | 22 | 19 | 10 | 7 | 31
  Day 29 | 9 | 30 | 34 | 9 | 30 | 37
  Day 36 | 28 | 37 | 33 | 39 | 37 | 37
  Day 43 | 38 | 38 | 32 | 41 | 40 | 37
  Day 50 | 34 | 39 | 30 | 41 | 37 | 36
  Day 64 | 27 | 39 | 27 | 41 | 35 | 35
  Day 85 | 17 | 39 | 23 | 41 | 32 | 35
  Day 181 | 4 | 26 | 12 | 27 | 8 | 19
  Day 394 | 0 | 13 | 7 | 7 | 3 | 17

14. Secondary Outcome: Seroconversion Based on TNA ED50, Defined as a ≥4-fold Increase Over Pre-vaccination Levels, or a ≥4-fold Increase Over the Lower Limit of Quantification (LLOQ) if the Pre-vaccination Value is Below the LLOQ
Description: The percentage of subjects obtaining seroconversion based on TNA ED50 antibody levels. Seroconversion represents the minimum intended effect of vaccination.
Time Frame: Days 8, 22, 29, 36, 43, 50, 64, 85, 181, and 394
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 41 | 39 | 41 | 41 | 42 | 38
Participants
  Day 8 | 0 | 0 | 0 | 0 | 0 | 0
  Day 22 | 1 | 22 | 20 | 11 | 6 | 32
  Day 29 | 8 | 30 | 34 | 10 | 29 | 36
  Day 36 | 29 | 37 | 34 | 40 | 38 | 37
  Day 43 | 37 | 38 | 32 | 41 | 41 | 37
  Day 50 | 34 | 39 | 31 | 41 | 37 | 36
  Day 64 | 29 | 39 | 32 | 41 | 36 | 36
  Day 85 | 15 | 38 | 22 | 40 | 31 | 32
  Day 181 | 3 | 24 | 8 | 25 | 7 | 18
  Day 394 | 0 | 12 | 8 | 7 | 3 | 13

15. Secondary Outcome: Seroconversion Based on ELISA Anti-PA IgG, Defined as a ≥4-fold Increase Over Pre-vaccination Levels, or a ≥4-fold Increase Over the Lower Limit of Quantification (LLOQ) if the Pre-vaccination Value is Below the LLOQ
Description: The percentage of subjects obtaining seroconversion based on ELISA anti-PA IgG antibody levels. Seroconversion represents the minimum intended effect of vaccination.
Time Frame: Days 8, 22, 29, 36, 43, 50, 64, 85, 181, and 394
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Age ≥ 66 Years: BioThrax (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
Number analyzed (Participants) | 41 | 39 | 41 | 41 | 42 | 38
Participants
  Day 8 | 0 | 0 | 0 | 0 | 0 | 0
  Day 22 | 2 | 22 | 20 | 8 | 12 | 33
  Day 29 | 16 | 31 | 38 | 9 | 36 | 37
  Day 36 | 33 | 37 | 37 | 38 | 39 | 37
  Day 43 | 39 | 38 | 36 | 41 | 41 | 36
  Day 50 | 38 | 39 | 36 | 41 | 40 | 36
  Day 64 | 31 | 39 | 34 | 41 | 38 | 36
  Day 85 | 23 | 39 | 25 | 41 | 32 | 28
  Day 181 | 4 | 23 | 4 | 24 | 10 | 7
  Day 394 | 0 | 4 | 0 | 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study vaccine through Day 394.
Groups:
- Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29): Participants dosed intramuscularly (IM) on Days 1 and 15 with 0.5 mL AV7909 and dosed IM on Day 29 with 0.5mL placebo
Arm/Group | Age ≥ 66 Years: BioThrax (Day1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/49 | 0/52 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/50 | 3/50 | 3/49 | 2/52 | 0/52 | 2/52
Other Adverse Events (participants affected / at risk) | 49/50 | 46/50 | 44/49 | 50/52 | 50/52 | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age ≥ 66 Years: BioThrax (Day1, Day 15, Day 29) (N=50) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) (N=50) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) (N=49) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) (N=52) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) (N=52) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) (N=52)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age ≥ 66 Years: BioThrax (Day1, Day 15, Day 29) (N=50) | Age ≥ 66 Years: AV7909 (Day 1, Day 15, Day 29) (N=50) | Age ≥ 66 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) (N=49) | Age ≥ 66 Years: AV7909 (Day 1, Day 29) With Placebo (Day 15) (N=52) | Age 18-50 Years: BioThrax (Day 1, Day 15, Day 29) (N=52) | Age 18-50 Years: AV7909 (Day 1, Day 15) With Placebo (Day 29) (N=52)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Chills (General disorders) | 0 (0) | 2 (4) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Fatigue (General disorders) | 9 (12) | 17 (25) | 14 (17) | 14 (21) | 10 (14) | 21 (28)
Injection site bruising (General disorders) | 12 (14) | 4 (4) | 7 (8) | 3 (4) | 9 (10) | 7 (7)
Injection site discolouration (General disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 34 (74) | 13 (18) | 7 (8) | 7 (8) | 27 (55) | 5 (5)
Injection site induration (General disorders) | 34 (74) | 15 (22) | 7 (7) | 11 (14) | 29 (57) | 12 (14)
Injection site mass (General disorders) | 38 (93) | 10 (12) | 5 (5) | 12 (16) | 37 (75) | 8 (9)
Injection site movement impairment (General disorders) | 7 (10) | 22 (31) | 10 (17) | 10 (13) | 15 (30) | 24 (32)
Injection site pain (General disorders) | 44 (152) | 41 (126) | 36 (77) | 43 (91) | 49 (191) | 50 (138)
Injection site pruritus (General disorders) | 26 (48) | 7 (9) | 3 (3) | 4 (6) | 30 (60) | 5 (7)
Injection site warmth (General disorders) | 26 (65) | 21 (31) | 11 (13) | 15 (25) | 27 (60) | 13 (19)
Pyrexia (General disorders) | 0 (0) | 3 (4) | 5 (5) | 5 (6) | 3 (3) | 7 (8)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (3) | 7 (8) | 5 (5) | 1 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 11 (19) | 8 (9) | 13 (20) | 8 (12) | 26 (37)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 11 (17) | 18 (41) | 6 (16) | 17 (26) | 12 (17) | 26 (37)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed. Data and results are owned by Sponsor. Results can be used by Institution for (a) internal non-commercial research, education and patient care, and (b) as required under applicable laws and regulations. Other uses require prior written consent of Sponsor.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT03518125/SAP_001.pdf
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT03518125/Prot_002.pdf